CLINICAL TRIAL: NCT07087873
Title: Assessment of Transcranial Alternating Current Stimulation's Clinical Efficacy in Treating Cognitive Impairment of Idiopathic Inflammatory Demyelinating Diseases
Acronym: TACS-CI-IIDDs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: [2025]086-002
Record Dates: First submitted 2025-06-24; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Inflammatory Demyelinating Disorders of the Central Nervous System; MS (Multiple Sclerosis); NMOSD; Acute Disseminated Encephalomyelitis; Transcranial Alternating Current Stimulation
MeSH Terms: conditions — Multiple Sclerosis; Encephalomyelitis, Acute Disseminated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromodulation group (Active Comparator)
  Interventions: Device: Neuroelectrical modulation group
- Pseudoneuromodulation group (Placebo Comparator)
  Interventions: Device: Pseudo-neuromodulation group

INTERVENTIONS:
Device: Neuroelectrical modulation group — Participants received transcranial electrical stimulation using the Spanish Neuroelectrics StarStim 32 device.
  Arms: Neuromodulation group
Device: Pseudo-neuromodulation group — Pseudo-stimulation is performed using the same equipment and procedures as in the neuromodulation group.
  Arms: Pseudoneuromodulation group

SUMMARY:
This study aims to explore the imaging and electrophysiological characteristics of idiopathic inflammatory demyelinating diseases (IIDDs), and their correlation with clinical manifestations. It also evaluates the effectiveness of transcranial electrical stimulation in alleviating clinical symptoms of IIDDs patients, and analyzes the key factors affecting the treatment efficacy. By uncovering the overall and individual characteristics of IIDDs, this study seeks to enhance therapeutic outcomes through personalized neuromodulation programs. The findings will provide a basis for applying non-invasive brain stimulation (NIBS) in IIDDs treatment and offer new ideas for future personalized medicine approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years old.
* Diagnosis: Patients with neuromyelitis optica spectrum disease, multiple sclerosis and other inflammatory demyelinating diseases of the central nervous system that meet the diagnostic criteria.
* Medications have been stable for at least three months.

Exclusion Criteria:

* Recurrence has been recorded in the past 3 months.
* Have a pacemaker or other metal implant in the body.
* Impaired skin integrity at the site of electrode placement.
* Previous organic brain disease such as epilepsy, hydrocephalus, central nervous system tumors, brain injury, or intracranial infection.
* Combined with severe or unstable organic diseases, such as heart, liver and kidney and other organ dysfunction.
* Pregnant or lactating women, those who are planning to become pregnant in the near future.
* Patient compliance is poor.
* In the opinion of the investigator, there is a situation that is not suitable to participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 128 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Expanded Disability Status Scale, EDSS score | At the 5-day point of treatment and 1 month following the end of treatment
  0-10 points, the higher the score, the more serious
Symbol Digit Modalities Test (SDMT) scale | At the 5-day point of treatment and 1 month following the end of treatment
  0-110 points, the higher the score, the better the cognitive function
Scoring results for tasks 1 and 7 in the Alzheimer disease assessment scale-cog(ADAS-cog) | At the 5-day point of treatment and 1 month following the end of treatment
  the higher the score, the better the cognitive function

SECONDARY OUTCOMES:
Mini-mental State Examination（MMSE） | At the 5-day point of treatment and 1 month following the end of treatment
  0-30，the higher the score, the better the cognitive function
Montreal-Cognitive Assessment（MoCA） | At the 5-day point of treatment and 1 month following the end of treatment
  0-30，the higher the score, the better the cognitive function
Stroop Color-Word Test score | At the 5-day point of treatment and 1 month following the end of treatment
  the higher the score, the better the cognitive function
Hamilton Depression Scale，HAMD | At the 5-day point of treatment and 1 month following the end of treatment
  The higher the score, the worse the depression.
Hamilton Anxiety Scale，HAMA | At the 5-day point of treatment and 1 month following the end of treatment
  The higher the score, the worse the anxiety.
a subjective questionnaire，adverse effects | Following the first day of treatment，Following the second day of treatment，Following the third day of treatment，Following the fourth day of treatment，Following the fifth day of treatment
  The intensity is scored from 0 to 4

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No